CLINICAL TRIAL: NCT04258930
Title: Randomized Comparative Open Trial of Occlusive Therapy With a Hydrocolloid or Silicone Versus Conventional Drying Treatment for the Local Care of Acute Lesions Caused by Herpes Zoster.
Brief Title: Occlusion vs Standard Treatment for the Treatment of Herpes Zoster
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Nacional para la Enseñanza y la Investigación de la Dermatología A.C. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNEIDAC-HZ-122-19
Record Dates: First submitted 2020-01-15; First posted 2020-02-06 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Aluminum Hydroxide; aluminum acetate; Bandages, Hydrocolloid

STUDY DESIGN:
Intervention Model Description: Randomized comparative open trial comparing occlusive therapy with hydrocolloid dressings versus a silicone gel vs a drying solution (standard care) to treat the rash of herpes zoster.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Aluminum sulphate and calcium acetate drying soaks (Active Comparator): Group A will receive 10 minute soaks every 8 hours with a solution prepared with aluminum sulphate and calcium acetate powder (Domeboro® (Advaita Pharmaceuticals, México)) diluted in 500 ml of clean cold water.
  Interventions: Other: Aluminum sulphate and calcium acetate drying soaks
- Group B: Topical sterile silicone gel for wounds (Experimental): Group B will receive topical silicone sterile gel for wounds (Stratamed gel®, (Stratapharma, Switzerland)) applied every 8 hours.
  Interventions: Device: Topical sterile silicone gel for wounds
- Group C: Hydrocolloid dressing (Experimental): Group C will apply an extra thin hydrocolloid dressing to all the open areas (Duoderm Extra Thin® (Convatec, USA)) with dressing changes every 48 to 72 hours depending on the amount of wound exudate.
  Interventions: Device: Hydrocolloid dressing

INTERVENTIONS:
Other: Aluminum sulphate and calcium acetate drying soaks — Dilute one envelope of the powder in 500 ml of clean cold water and apply for 10 minutes every 8 hours until completely healed.
  Other Names: Domeboro
  Arms: Group A: Aluminum sulphate and calcium acetate drying soaks
Device: Topical sterile silicone gel for wounds — Apply a thick layer of silicone gel to all open areas every 8 hours until completely healed.
  Other Names: Stratamed gel
  Arms: Group B: Topical sterile silicone gel for wounds
Device: Hydrocolloid dressing — Apply enough hydrocolloid dressings to cover all open areas and change every 2 to 3 days once the dressing becomes saturated (starts to drain around the borders).
  Other Names: Duoderm Extra-thin
  Arms: Group C: Hydrocolloid dressing

SUMMARY:
This study evaluates the addition of occlusive dressings (hydrocolloids) or topical silicone gel in the treatment of shingles (herpes zoster). One third of the participants will receive a hydrocolloid occlusive dressing, one third will receive the topical silicone gel and one third will receive the current treatment of the rash consisting of drying solutions (soaks).

DETAILED DESCRIPTION:
Herpes zoster (HZ), also known shingles, is a viral disease caused by the varicella-zoster virus. It is considered a local reactivation of varicella (chicken pox). The rash of herpes zoster is characterized by vesicles that appear following a single dermatome (the territory that is innervated by one spinal nerve). These vesicles may be very painful and cause discomfort due to draining and crusting. When a person becomes sick with shingles healthcare professionals prescribe systemic (oral) treatment with antivirals (e.g. acyclovir) and pain medication according to the type and severity. To treat the local lesions caused by shingles, over the centuries, patients have been treated with drying solutions and drying powders. This practice has been passed on through the years without any evidence supporting its effectiveness, in all likelihood due to the fact that the rash is self-limited to 2 to 3 weeks. Recently, new evidence has shown that the vesicles that appear with the shingles rash are not superficial but involve deeper areas of the skin and should be considered partial thickness wounds. Since 1962, it has become clear that partial thickness wounds benefit from occlusive therapy (keeping wounds closed and avoiding drying) such as dressings and occlusive gels that keep the wound wet rather than allowing it to dry.

In this clinical trial the investigators believe that given this information, using occlusive therapy with a hydrocolloid dressing or a silicone-based gel may heal the rash of herpes zoster, decrease pain and improve the quality of life, much faster than the treatment currently used of drying the area with powders and solutions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of HZ confirmed by a certified dermatologist
* Patients having maximum 72 hours from the start of the first vesicle
* Older than 18 years

Exclusion Criteria:

* Patients with dimethicone allergy
* Patients with hydrocolloid allergy
* Patients with acetaminophen allergy
* Patients with aluminium sulphate and calcium acetate allergy
* Patients with acyclovir allergy
* Pregnant women
* Breastfeeding women
* Unable to give informed consent
* Patients with signs of infection over the skin rash
* Patients with disseminated HZ
* Patients with hemorrhagic HZ
* Patients with complications such as pneumonia or encephalitis
* Patients unable to apply the treatment to the affected area
* Patients with HZ-associated keratitis
* Patients whose rash is located to hairy areas that may hinder occlusion with the hydrocolloid dressing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of days to achieve complete healing of cutaneous lesions. | Evaluation at 10 days.
  The total number of days from the beginning of the rash to the disappearance of all scabs.
Change in pain score using the Zoster Brief Pain Inventory (ZBPI) | Evaluation at baseline, 5 days, 10 days and 40 days.
  Score reduction in the Zoster Brief Pain Inventory (ZBPI). It uses an 11-point Likert scale (0-10) to rate herpes zoster pain and discomfort for four different dimensions (worst, least, and average during the past 24 hours, and now) and herpes zoster pain and discomfort-related interference with seven items of activities of daily living and health: general activity, mood, walking ability, work, relations with others, sleep, enjoyment of life.
Pain reduction as per acetaminophen need | Evaluation at 40 days.
  Amount of acetaminophen taken in total for pain control through the duration of the trial.
Change in the quality of life score as measured by the Dermatology Life Quality Index (DLQI) | Evaluation at baseline, 5 days, 10 days and 40 days.
  Quality of life score improvement as measured by the Dermatology Life Quality Index (DLQI). There are 10 questions, covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, treatment. Each question refers to the impact of the skin disease on the patient's life over the previous week. Each question is scored from 0 to 3, giving a possible score range form 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).

SECONDARY OUTCOMES:
Description and quantification of any side effect during the trial. | Evaluation at baseline, 5 days, 10 days and 40 days.
  Presence or absence of side effects of any of the above treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Contreras-Ruiz, MD, Principal Investigator — Fundación Nacional para la Enseñanza y la Investigación de la Dermatología A.C.
Locations (1):
- Hospital General Dr Manuel Gea González, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Boivin G, Jovey R, Elliott CT, Patrick DM. Management and prevention of herpes zoster: A Canadian perspective. Can J Infect Dis Med Microbiol. 2010 Spring;21(1):45-52. doi: 10.1155/2010/178036. PMID 21358885
- [Background] Bader MS. Herpes zoster: diagnostic, therapeutic, and preventive approaches. Postgrad Med. 2013 Sep;125(5):78-91. doi: 10.3810/pgm.2013.09.2703. PMID 24113666
- [Background] Cohen JI. Clinical practice: Herpes zoster. N Engl J Med. 2013 Jul 18;369(3):255-63. doi: 10.1056/NEJMcp1302674. PMID 23863052
- [Background] Coplan PM, Schmader K, Nikas A, Chan IS, Choo P, Levin MJ, Johnson G, Bauer M, Williams HM, Kaplan KM, Guess HA, Oxman MN. Development of a measure of the burden of pain due to herpes zoster and postherpetic neuralgia for prevention trials: adaptation of the brief pain inventory. J Pain. 2004 Aug;5(6):344-56. doi: 10.1016/j.jpain.2004.06.001. PMID 15336639
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Greenwood JE, Wagstaff MJ, Mackie IP, Mustoe TA. Silicone action in the open wound: a hypothesis. J Burn Care Res. 2012 Jan-Feb;33(1):e17-20. doi: 10.1097/BCR.0b013e31823e68cc. No abstract available. PMID 22138810
- [Background] HINMAN CD, MAIBACH H. EFFECT OF AIR EXPOSURE AND OCCLUSION ON EXPERIMENTAL HUMAN SKIN WOUNDS. Nature. 1963 Oct 26;200:377-8. doi: 10.1038/200377a0. No abstract available. PMID 14087904
- [Background] Karlsmark T, Goodman JJ, Drouault Y, Lufrano L, Pledger GW; Cold Sore Study Group. Randomized clinical study comparing Compeed cold sore patch to acyclovir cream 5% in the treatment of herpes simplex labialis. J Eur Acad Dermatol Venereol. 2008 Nov;22(10):1184-92. doi: 10.1111/j.1468-3083.2008.02761.x. Epub 2008 May 6. PMID 18462303
- [Background] Keegan DA. Reducing pain in acute herpes zoster with plain occlusive dressings: a case report. J Med Case Rep. 2015 Apr 25;9:89. doi: 10.1186/s13256-015-0560-5. PMID 25907451
- [Background] Lin PL, Fan SZ, Huang CH, Huang HH, Tsai MC, Lin CJ, Sun WZ. Analgesic effect of lidocaine patch 5% in the treatment of acute herpes zoster: a double-blind and vehicle-controlled study. Reg Anesth Pain Med. 2008 Jul-Aug;33(4):320-5. doi: 10.1016/j.rapm.2007.02.015. PMID 18675742
- [Background] Monk EC, Benedetto EA, Benedetto AV. Successful treatment of nonhealing scalp wounds using a silicone gel. Dermatol Surg. 2014 Jan;40(1):76-9. doi: 10.1111/dsu.12366. Epub 2013 Nov 25. No abstract available. PMID 24267314
- [Background] O'Brien L, Jones DJ. Silicone gel sheeting for preventing and treating hypertrophic and keloid scars. Cochrane Database Syst Rev. 2013 Sep 12;2013(9):CD003826. doi: 10.1002/14651858.CD003826.pub3. PMID 24030657
- [Background] Patel AR, Romanelli P, Roberts B, Kirsner RS. Treatment of herpes simplex virus infection: rationale for occlusion. Adv Skin Wound Care. 2007 Jul;20(7):408-12. doi: 10.1097/01.ASW.0000280199.58260.62. PMID 17620742
- [Background] Patel AR, Romanelli P, Roberts B, Kirsner RS. Herpes simplex virus: a histopathologic study of the depth of herpetic wounds. Int J Dermatol. 2009 Jan;48(1):36-40. doi: 10.1111/j.1365-4632.2009.03788.x. PMID 19126048
- [Background] Pott FS, Meier MJ, Stocco JG, Crozeta K, Ribas JD. The effectiveness of hydrocolloid dressings versus other dressings in the healing of pressure ulcers in adults and older adults: a systematic review and meta-analysis. Rev Lat Am Enfermagem. 2014 May-Jun;22(3):511-20. doi: 10.1590/0104-1169.3480.2445. PMID 25029065
- [Background] Tsai TF, Yao CA, Yu HS, Lan CC, Chao SC, Yang JH, Yang KC, Chen CY, White RR, Psaradellis E, Rampakakis E, Kawai K, Acosta CJ, Sampalis JS. Herpes zoster-associated severity and duration of pain, health-related quality of life, and healthcare utilization in Taiwan: a prospective observational study. Int J Dermatol. 2015;54(5):529-36. doi: 10.1111/ijd.12484. Epub 2014 Sep 10. PMID 25209019
- [Background] Uva L, Aphale AN, Kehdy J, Benedetto AV. Erosive pustular dermatosis successfully treated with a novel silicone gel. Int J Dermatol. 2016 Jan;55(1):89-91. doi: 10.1111/ijd.13066. Epub 2015 Sep 4. No abstract available. PMID 26341747
- [Background] WINTER GD. Formation of the scab and the rate of epithelization of superficial wounds in the skin of the young domestic pig. Nature. 1962 Jan 20;193:293-4. doi: 10.1038/193293a0. No abstract available. PMID 14007593
- [Background] Strauss SE, Oxman NM. Varicella and Herpes Zoster. In: Freedberg IM, Eisen AZ, Wolff K, Kopff A, et al. editors. Fitzpatrick´s dermatology in general medicine. New York, McGraw-Hill 1999, pp 2427-49.